CLINICAL TRIAL: NCT06467526
Title: Efficacy and Safety of Hydroxychloroquine in the Treatment of Sudden Sensorineural Hearing Loss
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRPG8P0011
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sudden Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Hydroxychloroquine; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine group (Experimental): Hydroxychloroquine with steroid
  Interventions: Drug: Hydroxychloroquine; Drug: Steroid
- Control group (Other): Steroid only
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral hydroxychloroquine (400mg/day) for 2 months
  Arms: Hydroxychloroquine group
Drug: Steroid — Oral prednisolone (5 mg) for 2 weeks (1 mg/kg/day for one week with gradually taper for another week with or without intratympanic dexamethasone 5 mg/ml injection for 2-4 times)

SUMMARY:
Sudden sensorineural hearing loss (SSNHL) is diagnosed when there's a sudden drop in hearing of at least 30 decibels across three consecutive frequencies, emerging within up to 72 hours. In clinical settings, steroids are the predominant treatment for SSNHL. However, the outcomes for patients undergoing steroid therapy for SSNHL can differ substantially. Moreover, a systematic review of randomized clinical trials has found no conclusive evidence pinpointing an effective treatment for SSNHL. Hydroxychloroquine, a derivative of chloroquine, is a medication that has gained attention for its potential role in modulating the immune response. We aim to see if hydroxychloroquine could augment hearing recovery in SSNHL under steroid treatment and to evaluate the safety of hydroxychloroquine in the treatment of SSNHL patients. We plan to enroll 80 SSNHL patients who received oral steroid therapy and randomize them into an experimental group (hydroxychloroquine with prednisolone, 40 patients) and a control group (prednisolone, 40 patients). The primary endpoint will be the change in pure tone audiogram (PTA) in the affected ear from screening until 3 months. The secondary endpoints will be the change in word recognition score and the change in bilateral tinnitus severity after treatment. Any side effects will be recorded to ensure the safety of this clinical trial.

DETAILED DESCRIPTION:
Sudden sensorineural hearing loss (SSNHL) significantly affects a patient's social and interpersonal interactions. It presents as an abrupt decrease in hearing, usually within a matter of hours or days. SSNHL typically impacts one ear and can range in severity, sometimes resulting in total deafness. In clinical settings, steroids are the predominant treatment for SSNHL. Yet, the outcomes for patients undergoing steroid therapy for SSNHL can differ substantially. Hydroxychloroquine, a derivative of chloroquine, is a medication that has gained attention for its potential role in modulating the immune response. Our study hypothesized that hydroxychloroquine could help the hearing recovery during the steroid treatment for SSNHL.

In this project, we will enroll two groups of subjects for our study.

1. Experimental group: Treatment with oral prednisolone (5 mg) for 14 days (high dosage 1 mg/kg/day for 7 days and gradually taper in the next week) and hydroxychloroquine for 60 days (400 mg/day)
2. Control group: Treatment with oral prednisolone (5 mg) for 14 days (high dosage 1 mg/kg/day for 7 days and gradually taper in the next week)

A. Primary endpoint:

The primary outcome measure for this study is the change in pure tone audiogram (PTA) in the affected ear from screening until 3 months. The PTA will be calculated as the arithmetic mean of air conduction thresholds at the frequency of 0.5k, 1k, 2k, and 4 kHz.

B. Secondary endpoints:

1. the change in PTA in the bilateral ear from screening until one week, two weeks, one month, and two months
2. change in word recognition score (WRS) in the bilateral ear from screening to one week, two weeks, one month, two months and three months
3. The grade of hearing recovery by Siegel's criteria from screening to 3 months
4. Percentage of recovery from screening until 3 months
5. change in bilateral tinnitus severity (evaluted by VAS and THI) from screening to one month, 2 months and 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral idiopathic sudden sensorineural hearing loss ≥ 30 dB in at least 3 consecutive frequencies, compared to the contralateral ear, within 3 days
2. Enrollment has to be accomplished within 14 days after SSNHL onset
3. Male or female aged ≥ 18 to 70 years
4. Ability to understand and follow the study protocol

Exclusion Criteria:

1. Pregnant or breast-feeding female
2. positive pregnancy test before receiving the study drug
3. Due to a history of physical efforts suspected perilymph fistula or membrane rupture.
4. Previously existing, known retrocochlear hearing loss
5. Any history of any ear operation or chronic inflammatory disease of middle ear in the past one year
6. History of blunt or penetrating ear trauma, head trauma, barotrauma, or acoustic trauma immediately preceding SSHL.
7. History of Meniere's disease, autoimmune hearing loss, radiation-induced hearing loss, endolymphatic hydrops, and otosclerosis.
8. History of chronic inflammatory diseases or autoimmune diseases
9. Prior chemotherapy or treatment with immunosuppressant drugs
10. Patients on renal dialysis
11. Patients with history of retinopathy, or are using drugs that could induce retinopathy, such as Tamoxifen
12. History of allergy to hydroxychloroquine
13. Patients who are contraindicated with oral steroid treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Hearing improvement | from screening until 3 months
  To evaluate if hydroxychloroquine could increase the hearing improvement

SECONDARY OUTCOMES:
Word recognition score | from screening until 3 months
  To evaluate if hydroxychloroquine could increase the word recognition score
Tinnitus severity | from screening until 3 months
  To evaluate if hydroxychloroquine could decrease the tinnitus severity

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Hui Yang, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No